CLINICAL TRIAL: NCT01888068
Title: Comparison of Bioimpedance Body Composition Device Measurements: Predicate (EFG®) Versus Candidate (Vitality Analyzer™)
Brief Title: Comparison of Bioimpedance Body Composition Device Measurements
Status: Completed | Type: Observational
Sponsor: IPGDx, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: IPGDx_Protocol1
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Self-declared Healthy Subjects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — None acquired or retained

GROUPS / COHORTS (1):
- No treatment

SUMMARY:
A new investigational device (BIA/Vitality Analyzer™) is being compared to a United States Food and Drug Approved 'predicate' reference device (EFG®) to demonstrate that they provide equivalent measurements of body fat. Both devices are "over-the-counter" bioimpedance body composition analyzers (estimate of body fat). These devices are classified as 'Not Significant Risk' devices; they do not expose you to any significant risks.

DETAILED DESCRIPTION:
You will be asked if you are 'healthy' to help the sub-investigator decide if you can be in the study. This is part of the "screening" process.

If you are 'healthy,' you will be asked to read and sign the informed consent documents and then enter into the study. The study Sub-investigator will ask your age, standing height and body weight. This information is used to describe the study participants. You will lie down on a flat surface/table; remove your shoes, socks and any jewelry. Four adhesive electrodes will be attached to your right hand and foot (two on each hand and foot), a small clip will then be connected to each electrode. A low level, radiofrequency alternating electrical current (425 microamps at 50 kilohertz) will be introduced into one pair (hand and foot) and the voltage across your body will be measured (other hand and foot). You will not feel the current being introduced into your body. While you remain on the table, the test will be repeated with a second bioimpedance device. The time required to complete these tests is about fifteen minutes. Participation in this study will depend upon if you are healthy and meet the specific study guidelines.

Screening for this study includes:

1. You are between the ages of 18 and 99 years old
2. You declare that you are healthy and do not have any known disease condition
3. You are not pregnant
4. You do not have an implanted electrical defibrillator
5. You do not have a pacemaker

The method for determining body impedance is based on the conduction of an applied electrical current in the organism. In biological structures, application of a constant low-level alternating current results in an impedance to the spread of the current that is frequency dependent. The living organism contains intra- and extracellular fluids that behave as electrical conductors and cell membranes that act as electrical condensers and are regarded as imperfect reactive elements. At low frequencies (-1 kHz) the current mainly passes through the extracellular fluids, whereas at higher frequencies (50-800 kHz), it penetrates the intra- and extracellular fluids. Thus body fluids and electrolytes are responsible for electrical conductance, which is the inverse of resistance, and cell membranes are involved in capacitance.

In biological systems, electrical conduction is related to water and ionic distribution in the conductor. Because fat-free mass, which includes the protein matrix of adipose tissue, contains virtually all the water and conducting electrolytes in the body, conductivity is far greater in the fat-free mass than the fat mass of the body. This hypothetical relationship was proposed by Nyboer et al., who demonstrated that electrically determined biological volumes (V) were inversely related to resistance (R), and reactance (Xc). Because the magnitude of reactance is small relative to resistance, and resistance is a better predictor of impedance than is reactance, the expression for V becomes: V = pL2/R, where R is in ohms.

ELIGIBILITY:
Inclusion Criteria:

* self-reported healthy men and women
* 18 to 99 years of age

Exclusion Criteria:

* Pregnancy
* Pacemaker
* Implanted Electrical Defibrillator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Self declared healthy subjects aged 18 to 99
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Comparison between the measured results of the candidate and predicate devices | One time thirty minute enrollment for two measurements
  Measured results from the candidate and predicate devices will be collected and compared

CONTACTS AND LOCATIONS:
Overall Officials: Hank C Lukaski, PhD, Principal Investigator
Locations (2):
- United States (2):
  - FL Arm, Nokomis, Florida
  - IPGDx, LLC, Harrisville, Michigan